CLINICAL TRIAL: NCT02798029
Title: A Phase II Study of the Efficacy, Safety, and Cost of Frameless Fractionated Stereotactic Radiation for Parenchymal Brain Metastases
Brief Title: Frameless Fractionated Stereotactic Radiation in Treating Patients With Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0874; NCI-2016-01180 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0874 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (FFSRT) (Experimental): Patients undergo FFSRT daily over 30 minutes for 3-5 days.
  Interventions: Radiation: Frameless Fractionated Stereotactic Radiation Therapy

INTERVENTIONS:
Radiation: Frameless Fractionated Stereotactic Radiation Therapy
  Other Names: FFSRT; Frameless SRT; FSRS

SUMMARY:
This phase II trial studies the safety and efficacy of frameless fractionated stereotactic radiation therapy for brain metastases. Frameless fractionated stereotactic radiosurgery is a specialized radiation therapy that delivers 3 to 5, high dose fractions of radiation directly to the brain lesions while sparing normal tissues.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy and safety of frameless fractionated stereotactic radiation therapy (FFSRT) on the treatment of solitary and oligometastatic brain metastases in the MD Anderson Houston Area Locations, MD Anderson Radiation Treatment Centers in New Mexico, MD Anderson affiliates and the main campus of MD Anderson, for patients unable or unwilling to undergo frame-based stereotactic radiosurgery (SRS).

SECONDARY OBJECTIVES:

I. To assess 6-month local control, intracranial progression-free survival and overall survival.

II. To collect data on charges and reimbursements of patients treated with FFSRT to compare those charges and reimbursements if the same patients had been treated with single-fraction, frame-based gamma knife SRS.

OUTLINE:

Patients undergo FFSRT daily over 30 minutes for 3-5 days.

After completion of study treatment, patients are followed up every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* All patients with 1-4 metastatic brain lesions who are considered eligible for single-fraction, frame-based SRS, who are unable or unwilling to undergo frame-based SRS
* One to 4 untreated metastatic brain lesions
* Each brain lesion must be less than or equal to 5 cm in diameter and not an optimal surgical candidate
* Patient must be able have a magnetic resonance imaging (MRI) of the brain for treatment planning
* Histologic confirmation of malignancy
* For patients of childbearing potential, non-pregnant state, confirmed by negative serum or urine beta-human chorionic gonadotropin (HCG) within (7) days of planned radiation treatment
* Glomerular filtration rate (GFR) adequate for intravenous (IV) contrast delivery for imaging
* No concurrent chemotherapy
* Patient may have had prior therapy for brain metastasis, including radiosurgery and surgical resection at the discretion of the treating physician however only new untreated lesions will be followed on protocol.

Exclusion Criteria:

* Five or more metastatic brain lesions
* Brain lesion(s) greater than 5 cm in diameter
* Lesion(s) involving the brainstem, optic chiasm or optic nerve(s)
* Patients unable to have IV contrast for computed tomography (CT) and MRI imaging
* Patient unable to have an MRI of the brain
* Patients willing to be treated with frame-based gamma knife SRS at MD Anderson main campus or MD Anderson at the Woodlands
* Positive pregnant status confirmed by serum or urine pregnancy test
* Primary small cell lung cancer, myeloma, lymphoma, leukemia, or other histologies not optimally treated with SRS
* Patients currently receiving chemotherapy/biologic/immunotherapy as these need to be held during FFSRT
* Prior whole brain radiotherapy or conventional external beam radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-08-08 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Incidence of lesion failure based on imagining assessments for each lesion | Up to 1 year
Rates of local control | Up to 1 year
Intracranial progression free survival (PFS) | From enrollment to either the first observation of progression disease in the brain or death due to any cause, assessed up to 1 year
  Will be summarized using the Kaplan-Meier method and the 50th percentile of the Kaplan-Meier distribution will determine the median intracranial PFS.
Overall survival (OS) | Up to 1 year
  Will be summarized using the Kaplan-Meier method and the 50th percentile of the Kaplan-Meier distribution will determine the median intracranial OS.
Cost data | Up to 1 year
  Will be summarized using descriptive statistics such as mean, median, standard deviation, and range. Comparisons in cost between treatment modalities will be evaluated using a paired t-test where each patient will serve as his or her own control to determine if the cost of frameless fractionated stereotactic radiation therapy (FFSRT) is comparable to standard treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chun, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Presbyterian Hospital, Albuquerque, New Mexico
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas